CLINICAL TRIAL: NCT06148012
Title: Investigation Of Marginal Bone Loss In Implants With Different Surface Properties And Geometric Designs: A Retrospective Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Mert Karabağ, PhD, Recep Tayyip Erdogan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RTEUOralandMaxilloFacialSurg
Record Dates: First submitted 2023-11-13; First posted 2023-11-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2023-11

CONDITIONS: Implant Infection; Peri-Implantitis; Bone Loss
Keywords: dental implant; marginal bone loss; peri-implantitis; fractal analysis
MeSH Terms: conditions — Peri-Implantitis; Bone Diseases, Metabolic | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RTEU Oral and Maxillofacial Surgery (Experimental)
  Interventions: Other: dental implant

INTERVENTIONS:
Other: dental implant — Digital panoramic radiographs taken during the patients' treatment periods (T0, T1) were used in the study. Measurements of marginal bone levels on radiographs were performed using the "Image J" software. The distance between the most coronal part of the implant neck and the most apical part of the defect caused by marginal bone loss was measured.
  Fractal analysis (FA) was conducted on panoramic radiographs (OPG) with a size of 2952x1435 pixels and a depth of 32 bits. FA on these radiographs at T0 and T1 times was performed using the box counting method determined by White and Rudolp with the ImageJ program(23).

SUMMARY:
Purpose: The aim of this study was to investigate the influence of surface characteristics and geometric design on marginal bone loss and bone quality in dental implants.

Materials and Methods: A total of 378 implants from 114 patients were evaluated in this study using panoramic and periapical radiographs. Implants were categorized into 19 subgroups according to the jaw where they were placed, length, diameter, surface preparation, type of prosthetic superstructure, and neck design. Radiological evaluations were conducted based on radiographs obtained at the time of implant placement and 3 months after prosthetic loading. After obtaining measurements of marginal bone loss and fractal analysis data, the significance of differences between groups was statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Implants with a minimum length of 8 mm
* Implants with a minimum diameter of 3.5 mm
* Availability of panoramic and periapical radiographs at T0 (immediately after surgery) and T1 (3 months after prosthetic loading).

Exclusion Criteria:

* Presence of a systemic condition hindering dental implant treatment and routine check-ups
* History of regular alcohol/tobacco use
* Presence of severe parafunctional habits (bruxism, etc.)
* Prior grafting procedures before dental implant placement
* Implant failure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss around different dental implants | 180 days
  Number of Participants: 114 Number of Dental Implants: 378
  Implants will be categorized into 19 subgroups according to the jaw where they were placed, length, diameter, surface preparation, type of prosthetic superstructure, and neck design. Radiological evaluations will be conducted based on radiographs obtained at the time of implant placement and 3 months after prosthetic loading.
  The distance between the most coronal part of the implant neck and the most apical part of the defect caused by marginal bone loss(millimeters) will be measured. The magnification ratio will be calculated by comparing the previously recorded implant length with the length measured on the software, allowing the determination of the actual value of MBL.
Fractal values around dental implant radiographs | 180 days
  A total of 378 implants from 114 patients will be evaluated in this study using panoramic and periapical radiographs. Implants will be categorized into 19 subgroups according to the jaw where they were placed, length, diameter, surface preparation, type of prosthetic superstructure, and neck design. Radiological evaluations will be conducted based on radiographs obtained at the time of implant placement and 3 months after prosthetic loading. And measurement pre op post op fractal values

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University Oral an Mazillofacial Surgery, Rize, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No